CLINICAL TRIAL: NCT05739760
Title: Cuddle-Calm Booklets - Increasing Mother-child Emotional Connection Through the Use of a Nurture-based Children's Book
Brief Title: Impact of Cuddle and Calm Booklets on Parent-Child Emotional Connection a Nurture-based Children's Book
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Student research, student left the university
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G Welch, Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology) at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAT2041
Record Dates: First submitted 2021-04-14; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Emotional Problem
MeSH Terms: interventions — Safety; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families assigned the "Cuddle and Calm" booklet (Experimental): A poem about emotional expression in times of upset
  Interventions: Behavioral: Poem book about relational health
- Families assigned the "Health and Safety" booklet (Experimental): A poem about health and safety with tips on topics such as first aid and injury prevention
  Interventions: Behavioral: Poem book about physical health and safety

INTERVENTIONS:
Behavioral: Poem book about relational health — Poem book will consist of illustrations, poetry, and tips for parents on how to resolve their child's upset, their own upset, and to develop a stronger relationship. The study physician may read the book to the families at the visit. Then, families are instructed to read the book at least once, for as many times as the parent opts to.
  Other Names: "Cuddle and Calm" booklet
  Arms: Families assigned the "Cuddle and Calm" booklet
Behavioral: Poem book about physical health and safety — Poem book will consist of illustrations, poetry, and tips for parents on how to keep their child physically healthy and safe, and to avoid accidental injuries. The study physician may read the book to the families at the visit. Then families are instructed to read the book at least once, for as many times as the parent opts to.
  Other Names: "Health and Safety" booklet
  Arms: Families assigned the "Health and Safety" booklet

SUMMARY:
Children's social and emotional development is affected by their relationship with their parents. The goal of the study is to test an intervention that guides parents and children to strengthen their relational health and navigate difficult situations. This study will begin in the well-child visit in the pediatric department at MetroHealth Medical Center. Pediatricians will invite families to enroll in the study, then study personnel will administer two illustrated poem books called "Cuddle and Calm," a poetry book with tips on how to strengthen the parent-child relationship, or "Health and Safety," a poetry book with tips on how to avoid injuries. This intervention is based on the construct of emotional connection as studied by Martha G Welch MD, who developed the Welch Emotional Connection Screen (WECS) along with Amie Hane PhD. The WECS-Parent Report (WECS-PR) is a likert scale parent-report screen with items regarding the domains featured in the WECS.

DETAILED DESCRIPTION:
The parent-child relationship affects the child's socio-emotional development and the parent's stress. The purpose of this study is to test a behavioral intervention designed to guide parents and children on how to strengthen their relational health and navigate challenging interactions. This intervention will involve a unique experience in the well-child visit in the pediatric department (either virtually or in-person) at Metrohealth Medical Center, in which pediatricians will invite families to participate in the study. Then, study personnel will administer either "Cuddle and Calm," an illustrated poetry book that feature tips on how to promote the relationship between parents and their children, or "Health and Safety," an illustrated poetry book that features tips on how to navigate risky injuries. The approach is based on the construct of emotional connection as studied by Dr. Martha Welch's Nurture Science Program of Columbia University Irving Medical Center. They developed the Welch Emotional Connection Screen (WECS), an assessment that allows parent-facing professionals to rate the emotional connection of a mother-child relationship in just a few minutes of observed interaction, and shows preliminary predictive properties when performed in the first year of life. The WECS-Parent Report (WECSPR) is a Likert-scale parent-report screen with items regarding the domains featured in the WECS. All consenting subjects will complete WECS-PR, a tantrum survey before and after administration of the booklets to determine the impact of the reading material.

ELIGIBILITY:
Inclusion Criteria:

* Children between 18 months and 6 years old and their mothers or grandmothers, if primary caregiver, scheduled for a well visit.

Exclusion Criteria:

* Refusal to consent
* Inability to access internet; not having an email address.

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
Change in Tantrum Questionnaire Score | Change from baseline to 4 weeks post book reading
  Determine whether mother-child dyads who received "Cuddle and Calm," had better scores on the tantrum questionnaire compared to the dyads who received the control book poem books, "Health and Safety."

SECONDARY OUTCOMES:
Welch Emotional Connection Screen - Parent Report | change from baseline to 4 weeks post book reading
  Test the effect of "Cuddles and Calm" on emotional connection operationalized as the Welch Emotional Connection Screen - Parent Report

OTHER OUTCOMES:
Book Acceptability Questionnaire Score | 4 weeks after receiving designated books
  Assess acceptability of the poem booklets through Likert-scale questions about liking the books. This is a 11-item questionnaire with a score range of 11 to 55. 11 = low acceptability and 55 = high acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology)